CLINICAL TRIAL: NCT04043728
Title: Addressing Psychological Risk Factors Underlying Smoking Persistence in COPD Patients: The Fresh Start Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORA # 18082201
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Copd; Smoking Cessation; Nicotine Dependence; Tobacco Use; Cigarette Smoking
Keywords: COPD; Smoking cessation; Nicotine dependence; Tobacco use; Cigarette smoking; Behavioral treatment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking Cessation; Tobacco Use Disorder; Tobacco Use; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness (Experimental): This module introduces mindfulness training skills, with the goal of cultivating nonjudgmental, present-focused experience of emotions, thoughts, and physical sensations related to cigarette smoking. By progressing though a series of experiential exercises (e.g., awareness of the breath, anchoring in the present), this module seeks to reduce maladaptive attempts to control negative emotions and facilitate tolerance of the physical and emotional symptoms of nicotine withdrawal.
  Interventions: Behavioral: Unified Protocol adapted for smoking cessation
- Interoceptive Exposure (Practice Quitting) (Experimental): This module introduces interoceptive exposure, a technique in which participants purposefully and systematically complete exercises to evoke physical sensations typically associated with anxiety and distress, in order to reduce fear and avoidance of these sensations. Interoceptive exercises will focus on a gradual exposure to nicotine withdrawal symptoms, through a series of 'practice quit attempts' (i.e., brief periods of smoking abstinence without intention to permanently quit).
  Interventions: Behavioral: Unified Protocol adapted for smoking cessation
- Behavioral Activation (Countering Emotional Behaviors) (Experimental): This module introduces behavioral activation, which seeks to increase positive emotions by systematically introducing greater engagement with natural rewards. Treatment sessions focus on the identification of avoidance strategies, including cigarette smoking as a coping strategy for negative emotions. The goal of this treatment module is to replace smoking with adaptive coping strategies to facilitate contact with and enjoyment of reinforcing activities that are incompatible with smoking.
  Interventions: Behavioral: Unified Protocol adapted for smoking cessation

INTERVENTIONS:
Behavioral: Unified Protocol adapted for smoking cessation — Treatment components are cognitive-behavioral strategies adapted from the Unified Protocol (UP) for the Transdiagnostic Treatment of Emotional Disorders. Behavioral counseling strategies for smoking cessation, drawn from current US Public Health Service guidelines, are incorporated in each treatment module. All participants will be provided with the American Lung Association Freedom from Smoking guide to aid in their quit attempt.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is caused primarily by smoking and smoking cessation is the first-line treatment for slowing disease progression. Despite this, nearly 50% of COPD patients continue to smoke following diagnosis. Smokers with COPD report high rates of co-occurring conditions - nicotine dependence, depression, and anxiety - which serve as barriers to quitting. The current study will pilot test a behavioral intervention designed to target the common psychological factors underlying these co-occurring conditions and foster smoking cessation among COPD patients.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is caused primarily by smoking and smoking cessation is the first-line treatment for slowing disease progression. Despite this, nearly 50% of COPD patients continue to smoke following diagnosis. Smokers with COPD report high rates of co-occurring conditions - nicotine dependence, depression, and anxiety - which serve as barriers to quitting. The current study will pilot test a behavioral intervention designed to target the common psychological factors underlying these co-occurring conditions and foster smoking cessation among COPD patients. The specific aim is to:

Aim: Develop a multi-component behavioral treatment to address psychological risk factors among COPD patients. We will conduct a component analysis using single case design experiments with 15 participants to a) examine the contribution of each treatment component to the behavioral target of smoking for affect regulation, and b) establish proof-of-concept on the clinical endpoint of initial cessation (>24 hours abstinence).

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be males and females who are:

* Diagnosed with COPD (as documented in electronic health record [EHR]),
* Daily cigarette smokers (5 or more cigarettes per day over past 30 days),
* Intend to quit smoking within the next 60 days,
* Report at least moderate level of smoking for affective regulation (SMQ-R coping subscale score 30 or greater),
* Have access to a smart phone, tablet, or computer, and
* Are able to communicate fluently in English

Exclusion Criteria:

* Any concurrent medical or psychiatric condition which would preclude ability to provide informed consent or perform study procedures (e.g., moderate to severe dementia and/or severe, uncontrolled schizophrenia), as determined by the treating physician or study PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda R Mathew, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mathew AR, Avery EF, Cox C, Nwanah P, Kalhan R, Hitsman B, Powell LH. Development of a targeted behavioral treatment for smoking cessation among individuals with Chronic Obstructive Pulmonary Disease. J Behav Med. 2023 Dec;46(6):1010-1022. doi: 10.1007/s10865-023-00411-z. Epub 2023 May 6. PMID 37148395

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness | Interoceptive Exposure (Practice Quitting) | Behavioral Activation (Countering Emotional Behaviors)
Started | 6 | 6 | 6
Completed | 5 | 4 | 6
Not Completed | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness | Interoceptive Exposure (Practice Quitting) | Behavioral Activation (Countering Emotional Behaviors) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (6.1) | 61.5 (6.4) | 63.3 (4.0) | 60.6 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 14
  Male | 0 | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 6 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 6 | 16
  White | 1 | 1 | 0 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved 24-hour Smoking Abstinence at End-of-treatment
Description: The clinical endpoint will be achievement of 24-hour smoking abstinence at end-of-treatment, as verified by CO < 5 ppm.
Time Frame: 24 hours post-quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness | Interoceptive Exposure (Practice Quitting) | Behavioral Activation (Countering Emotional Behaviors)
Number analyzed (Participants) | 6 | 6 | 6
Participants | 1 | 1 | 2

2. Secondary Outcome: Percent Change in Smoking Motives Questionnaire-Revised (SMQ-R) Average Score
Description: The secondary outcome is percent change in Smoking Motives Questionnaire-Revised (SMQ-R) average score. The SMQ-R measures the construct of smoking for affect regulation (i.e., smoking to improve mood or reduce distress). SMQ-R average score is computed as the average of 13 items, each assessed on a 0 to 100 scale, with higher scores indicating greater smoking for affect regulation.
Time Frame: Through active treatment phase (approximately 4 weeks)
Measure: Mean (Standard Deviation); unit: Percent score change
Arm/Group | Mindfulness | Interoceptive Exposure (Practice Quitting) | Behavioral Activation (Countering Emotional Behaviors)
Number analyzed (Participants) | 6 | 6 | 6
Percent score change | -0.11 (0.24) | -0.32 (0.25) | -0.11 (0.20)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed over the course of active study participation (approximately 35-50 days).
Arm/Group | Mindfulness | Interoceptive Exposure (Practice Quitting) | Behavioral Activation (Countering Emotional Behaviors)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT04043728/Prot_SAP_000.pdf